CLINICAL TRIAL: NCT02853916
Title: Efficacy of a Brown Seaweed Powder for Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: innoVactiv Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2016:51
Record Dates: First submitted 2016-07-14; First posted 2016-08-03 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Blood Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 500 mg InSea2® (Active Comparator)
  Interventions: Dietary Supplement: 500 mg InSea2®
- 250 mg InSea2® (Active Comparator)
  Interventions: Dietary Supplement: 250 mg InSea2®
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 500 mg InSea2®
  Arms: 500 mg InSea2®
Dietary Supplement: 250 mg InSea2®
  Arms: 250 mg InSea2®
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The objectives of this trial are to confirm efficacy in human of a brown seaweed powder and explore dose-response relationship by comparing two different doses.

The primary endpoint is incremental area under the curve (iAUC, mmol*min/L) for blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged between 18-45 y
* Normoglycemic (fasting blood glucose <5.6 mmol/L)
* Body mass index (BMI) 18.5-29.9 kg/m2
* Able to consume bread products

Exclusion Criteria

* Fasting blood glucose > 5.6 mmol/L
* Systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg
* Previous history of cardiovascular disease, diabetes, liver or kidney disease, inflammatory bowel disease, celiac disease, short bowel syndrome, any malabsorptive syndrome, pancreatitis, gallbladder or biliary disease
* Presence of a gastrointestinal disorder within the past year
* Presence of major gastrointestinal surgeries
* Thyroid problems
* Smokers
* Consuming prescription or non-prescription drug, herbal or nutritional supplements known to affect blood glucose or that could affect the outcome of the study as per investigator's judgement
* Women that are currently pregnant or lactating, or not using an appropriate contraception method
* Excessive alcohol intake (more than 2 drinks per day or more than 9 drinks per week)
* Allergic to shellfish (crab) or molluscs
* Weight gain or loss of at least 10lbs in previous three months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-08; Primary Completion 2017-04 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Incremental area under the curve (iAUC, mmol*min/L) of blood glucose | 0, 15, 30, 45, 60, 75, 90, 120, 150, 180 and 210 min
  Incremental area under the curve (iAUC, mmol*min/L)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Jones, PhD, Principal Investigator — University of Manitoba
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada